CLINICAL TRIAL: NCT07345416
Title: A Randomized, Single-Masked, Active-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of ST-1 Silicone Hydrogel Daily Disposable Soft Contact Lenses Compared to Miru 1day UpSide
Brief Title: A Clinical Trial Assessing the Efficacy and Safety of ST-1 Silicone Hydrogel Daily Disposable Soft Contact Lenses Compared to Miru 1day UpSide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STCT-01
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Myopia; Soft Contact Lenses; Daily Disposable Soft Contact Lenses
Keywords: Myopia; Soft Contact Lenses; Daily Disposable Soft Contact Lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and evaluators will be masked to the treatment assignment of the randomization code. Each site must have an unmasked staff member who will be responsible for dispensing and collecting the study test and control lenses. The randomization code will be provided to this unmasked staff member at the time of subject randomization.
  Although this design involves masking of both investigators and evaluators, the official protocol title refers to the study as "Single-Masked" because the subjects are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ST-1 (Experimental): Subjects will be randomized at Visit 1 with a 2:1 allocation ratio (approximately two-thirds assigned to this arm).
  Interventions: Device: ST-1
- Miru 1day UpSide (Active Comparator): Subjects will be randomized at Visit 1 with a 2:1 allocation ratio (approximately one-third assigned to this arm).
  Interventions: Device: Miru 1day UpSide

INTERVENTIONS:
Device: ST-1 — ST-1 lens worn in daily wear, daily disposable mode.
  Arms: ST-1
Device: Miru 1day UpSide — Miru 1day UpSide lens worn in daily wear, daily disposable mode.
  Arms: Miru 1day UpSide

SUMMARY:
This study will enroll 63 eligible subjects (126 eligible eyes, complete at least 108 evaluable eyes) in approximately 6 different medical centers in Taiwan, in order to evaluate the efficacy and safety of ST-1 silicone hydrogel daily disposable soft contact lenses (ST-1 lenses) compared to Miru 1day UpSide. Enrolled subjects will be randomized in a 2:1 test to control ratio at Visit 1. Each site will enroll 8 (intended minimum) to 12 (intended maximum) subjects. In order to eliminate the bias, the Investigators and the evaluators will be masked to the treatment assignment of the randomization code. During the study, the Investigator(s) will examine the ocular health via inquiry, slit lamp biomicroscopy (SLB), visual acuity (VA) test, keratometry, and refractive changes. The Investigator(s) will check ocular health and evaluate the inclusion/exclusion criteria of subjects at screening. After entering the study, subjects will be required to wear the lenses on a daily basis, record daily wearing time on a diary, return to the study site at scheduled visits for evaluations and complete the self-assessment questionnaire at Visit 2 to Visit 7 (1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged between 18 to 40 (inclusive) years old.
2. Diagnosis of myopia in both eyes, each ranging from -0.50D to 6.00D with manifest astigmatism of ≤ 1.00D per eye.
3. Understands and signs an informed consent form (ICF).
4. Willing to adhere to the instructions set forth in this study as well as understand and complete all specified evaluation.
5. Willing and able to refrain from using any other contact lenses other than those provided for the duration of the study.
6. Has experience and capability of wearing soft contact lenses.
7. Be a habitual soft contact lenses wearer in both eyes, defined as wearing lenses for at least 8 hours per day, 5 days per week, for a minimum duration of 30 days.
8. Tear breakup time (TBUT) > 5 seconds in each eye.

Exclusion Criteria:

1. Eyes with abnormality or disease as follows:

   1. Evidence of lid abnormality or infection (e.g., entropion, ectropion, chalazia, and recurrent styes).
   2. Clinically significant slit lamp findings (e.g., infiltrates or other slit lamp findings Level 2 or above: corneal edema, tarsal abnormalities, and conjunctival injection).
   3. Other active ocular disease (e.g., uveitis, corneal epithelial defect, severe dry eye, lacrimal duct defect, glaucoma, cornea [infiltrates], conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology).
   4. History of recurrent corneal erosions.
   5. Aphakia.
2. Ocular or systemic allergies or diseases that may interfere with contact lens wear, occur within 2 weeks prior to the Screening Visit.
3. Use of topical ocular medications, except artificial tear, within 7 days prior to the Screening Visit.
4. History of refractive, ocular, or intraocular surgery.
5. Participation in any clinical trial (with the exception of retrospectives studies) within 30 days prior to the Screening Visit.
6. Have risks in dangerous and significant eye edema, congestions, corneal abrasion or neovascularization when wearing contact lens.
7. Any corneal surface roughness.
8. Unable to achieve best corrected visual acuity (BCVA) of logMAR 0.1 or better in each eye at distance using manifest refraction.
9. Females who are pregnant, breastfeeding or who intend to become pregnant over the course of the study.
10. Current drug or alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirement.
11. Allergy to any component in the study product.
12. Subjects who wore monovision, multifocal, toric, or rigid contact lenses within 30 days prior to the Screening Visit.

    Note: Monovision is defined as a vision correction method for treating presbyopia in which the dominant eye is corrected for distance vision and the non-dominant eye is corrected for near vision.
13. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lenses wear at the Investigators discretion within 14 days prior to the Screening Visit.
14. Other conditions not suitable for participating in this study judged by the Investigators.
15. Live in dusty or pharmaceutical environments.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Corrected distance Logarithm of the Minimum Angle of Resolution (logMAR) visual acuity at the final visit (Visit 7) | Screening, 3 months following enrolment
  Assessed using a Tumbling E Series ETDRS® chart.

SECONDARY OUTCOMES:
Self-assessment of eye symptoms | Screening, 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  This questionnaire includes 11 items assessing symptoms during contact lens wear: discomfort, tearing, photophobia, itching, burning, halos, dryness, variable vision, blurred vision, pain, and other (specify if present).
  Scale: 0-4 (minimum = 0, maximum = 4), where higher scores indicate worse symptoms.
  Grades:
  0 = None
  1. = Trace
  2. = Mild
  3. = Moderate
  4. = Severe
Self-assessment of lens performance | Screening, 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  This questionnaire includes 5 items assessing lens performance during contact lens wear: insertion comfort, overall comfort, vision, insertion handling, and removal handling.
  Scale: 0-5 (minimum = 0, maximum = 5), where higher scores indicate worse performance.
  Grades:
  【comfort】 0 = Excellent
  1 = Very comfortable 2 = Comfortable 3 = Slightly uncomfortable 4 = Very uncomfortable 5 = Causes pain 【vision】 0 = Excellent
  1. = Very good
  2. = Good
  3. = Poor
  4. = Very poor
  5. = Unacceptable 【handling】
  0 = Excellent
  1. = Very good
  2. = Good
  3. = Poor
  4. = Very poor
  5. = Unmanageable
Total wearing hours | Daily for 3 months after enrollment
  Cumulative duration of lens wear throughout the study period, determined from the daily wearing time recorded by participants in the electronic patient-reported outcome (ePRO) diary.
Total wearing days | Daily for 3 months after enrollment
  Total number of days the study lenses were worn for 8 hours or more, based on the daily wearing time entered by participants in the electronic patient-reported outcome (ePRO) diary. A wearing day is defined as a day with 8 hours or more of lens wear.
Average wearing hour each time | Daily for 3 months after enrollment
  Average duration of lens wear for each individual application, derived from the wearing data entered by participants in the electronic patient-reported outcome (ePRO) diary.
Daily wearing hour | Daily for 3 months after enrollment
  Average number of hours the study lenses were worn per day, as recorded by participants in the electronic patient-reported outcome (ePRO) diary.
Corrected distance visual acuity (CDVA) change with the dispensed lenses from baseline | Screening, 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  Assessed using a Tumbling E Series ETDRS® chart.
Slit lamp biomicroscopy (SLB) findings | Screening, 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  Assessed using a slit lamp.
Change from baseline in keratometry readings | Screening, 3 months following enrolment
  To evaluate the absolute change from baseline in keratometry readings between Screening and the 3 months visit.
Percent change from baseline in keratometry readings | Screening, 3 months following enrolment
  To evaluate the percent change from baseline in keratometry readings between Screening and the 3-month visit.
Change from baseline in refractive parameters | Screening, 3 months following enrolment
  To evaluate the absolute change from baseline in refractive parameters, including sphere (S), cylinder (C), and axis (A), measured by subjective refraction test between Screening and the 3-month visit.
Percent change from baseline in refractive parameters | Screening, 3 months following enrolment
  To evaluate the percent change from baseline in refractive parameters, including sphere (S), cylinder (C), and axis (A), measured by subjective refraction test between Screening and the 3-month visit.
Adverse events | Screening, 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  AE will be evaluated by the investigator.
Lens fitting and surface assessment | 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  Lens fitting will be assessed with a slit lamp, and surface assessment will be assessed with a slit lamp or a stereomicroscope.
Device deficiency | 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months following enrolment
  A device deficiency refers to any inadequacy of the investigational product regarding identity, quality, durability, reliability, safety, or performance, including malfunctions, use errors, and labeling issues.
  Categories include:
  Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color) Lens cloudy or surface/edge defect Torn lens during handling/in pack Packaging deficit (e.g., mislabeled product, tampered seal, leaking container) Suspect contamination Lack of performance (e.g., fit changes under hypobaric or low-humidity conditions) Other
  If such an event occurs, investigators must evaluate, record, and report all deficiencies and malfunctions during the trial using the device deficiency evaluation form.
  The frequency of device deficiencies will be summarized for safety evaluation and compared between treatments.
Overall lens dicontinuation rate | Daily for 3 months after enrollment
  Permanent discontinuation of lens wear, if it occurs, will be recorded via ePRO. The overall discontinuation rate will be calculated and compared between treatments using Chi-square or Fisher's exact test.
Lens discontinuation rate by reason | Daily for 3 months after enrollment
  Reasons for permanent discontinuation (e.g., discomfort, adverse event, convenience), if they occur, will be collected via ePRO, categorized, and tabulated by visit and overall.
Lens replacement | Daily for 3 months after enrollment
  Lens replacement is defined as removal and reapplication of a lens, regardless of whether a new lens is used. If it occurs, all reasons (e.g., sleeping, rest, device deficiency, adverse events, other) will be recorded via ePRO and tabulated by visit and overall.
Artificial tears usage frequency | Daily for 3 months after enrollment
  Participants will record their daily usage of artificial tears via ePRO, if applicable. The record will include both the frequency of use and the number of drops applied each time.

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Changhua Christian Hospital, Changhua, Changhua City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City, New Taipei City
  - Taipei Veterans General Hospital, Taipei, Taipei City
  - Tri-Service General Hospital, Taipei, Taipei City
  - Chang-Gung Memorial Hospital LinKou Branch, Taoyuan District, Taoyuan City

IPD SHARING:
Plan to Share IPD: No